CLINICAL TRIAL: NCT04658953
Title: Comparison of the Effectiveness of Ultrasound-guided Versus Radioguided Medial Lumbar Bundle Branch Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Hôpital de Braine-l'Alleud (Other); Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE/20-11-10
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Low-back Pain; Lumbar Facet Joint Syndrome
Keywords: Pain; Fluoroscopy; Ultrasound; Injection Site Infiltration; Chronic; Lumbar facet joint syndrome; Medial branch blocks; Disability; Local anesthetic; Lumbalgia; Lumbar zygapophysial joint; Facet syndrome; Chronic Low-back Pain; Medial branch block
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided infiltration (Experimental): The patient is positioned in the prone position with a block under his stomach. After disinfection of the lumbosacral region with alcoholic chlorhexidine 0.5%, the investigators position the convex probe of the ultrasound machine in the transverse plane. Once the spine has been located, the investigators look for the spinous processes of the lower lumbar vertebrae L4 and L5 with the mark on the cranial side and the side opposite the mark on the side of the sacrum. The latter is visualized as a continuous hyperechoic line. Then, the probe is tilted 90 ° to be in a transverse plane. A 22G needle is introduced in a transverse axis starting from the laterality by inserting it in the direction of the median bone contacts of the lower lumbar vertebrae L3, L4 and L5. An infiltration will be unilaterally performed at three levels (L3-L4, L4-L5 and L5-S1 levels).
  Interventions: Other: Ultrasound guided infiltration
- Fluoroscopy-guided infiltration (Experimental): The patient is positioned in the prone position with a block under his stomach. The lumbosacral region is disinfected with alcoholic chlorhexidine 0.5%.
  The C-shaped arm of a X-ray fluoroscopy is positioned around the patient in an antero-posterior view tilted ¾ in order to free the classic view called "scotty dogs ". The puncture point is determined by the positioning of the needle in so-called "tunnel vision". The needle is thus brought to the bone contact corresponding to the eye of the scotty dog in tunnel vision, an area corresponding to the passage of the lumbar median branch. An infiltration will be unilaterally performed at three levels (L3-L4, L4-L5 and L5-S1 levels).
  Interventions: Other: Fluoroscopy guided infiltration

INTERVENTIONS:
Other: Ultrasound guided infiltration — In the patient in prone position, an infiltration guided by ultrasound will be performed in three puncture points (L3-L4, L4-L5 and L5-S1 levels unilaterally). At each level, 1mL of a mixture consisting of 3mL of Linisol 2% (60mg of lidocaine) and 1mL of Depomedrol 40mg / Lidocaine 10mg is injected.
  Arms: Ultrasound-guided infiltration
Other: Fluoroscopy guided infiltration — In the patient in prone position, an infiltration guided by fluoroscopy will be performed in three puncture points (L3-L4, L4-L5 and L5-S1 levels unilaterally). At each level, 1mL of a mixture consisting of 3mL of Linisol 2% (60mg of lidocaine) and 1mL of Depomedrol 40mg / Lidocaine 10mg is injected.
  Arms: Fluoroscopy-guided infiltration

SUMMARY:
In adults with chronic low back pain, the investigators will compare the effectiveness of the medial bundle branch block on three lumbar levels (L3-L4, L4-L5 and L5-S1) performed either by radiographic guidance or by ultrasound approach according to a transverse approach.

The objective of this study will be to evaluate the benefit of these both procedures on pain, on the practice of daily activities and the incidence of adverse events in order to show whether the two modalities are equivalent.

DETAILED DESCRIPTION:
"Lumbar facet syndrome" is a source of spinal distress affecting up to 45% of patients with chronic low back pain due to inflammation, degenerative or arthritic changes, overloading of the posterior or posterior lumbar facet joints.

First-line treatment for the relief of chronic low back pain of zygapophyseal joint origin includes bed rest, oral pain relievers / anti-inflammatory drugs, and physiotherapy. If unsuccessful, intra-articular injections and medial bundle branch block (BBM) provide diagnosis and are an alternative to neurotomy (radiofrequency or cryoneurolysis).

The BBM targets the medial branches of the posterior twigs, that is, it blocks the nociceptors and the muscles of the dermatome undertaken by targeting the medial branches of the dorsal vertebral branch supplying a facet above and below the vertebrae which ensure sensory innervation of the facet joint. The current standard technique is radiography requiring three punctures (transverse-axial plane) and the ultrasound technique is also described in this plan and also requires three puncture points. The investigatorswould like to compare this promising new technique to the standard radiographic technique since it would avoid irradiation and is easier to handle.

For this study, the investigatorswill compare the BBM on three lumbar levels (L3-L4, L4-L5 and L5-S1) performed under radiography versus ultrasound according to a transverse approach.

To compare the equivalence of this two modalities the investigators will evaluate :

* the benefit of the procedure on pain (via the visual analogue scale (VAS) collected before then at 1 week and at 1 month after the infiltrations)
* the evolution of the possibility of carrying out daily activities (via the Duke's activity status index (DASI) scale, collected at the same intervals as the VAS)
* the limits of daily activities (via the Oswestry Disability Index (ODI), collected at the same time intervals)
* the incidence of adverse events

A screening for anxiety and depressive disorders will be also performed before infiltration by the Hospital Anxiety and depression scale (HADS) comprising 14 items.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low-back pain for at least 3 months, without response to a conservative treatment of minimum 4 weeks
* No signs of dissociated pain, radiculitis, neurological diseases (including stroke, Parkinson's disease), spinal instability or deformities (such as scoliosis, ankylosing spondylitis), history of lumbar surgery , fracture or lumbar tumor.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Allergy to injected products (Depomedrol or Linisol)
* Psychiatric disorders hindering understanding of the protocol
* Local or systemic infection
* Coagulation disorder
* Obese with a BMI> 35 kg / m²

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) score | 1 month
  Change in Oswestry Disability Index (ODI) score from baseline to 1 month after infiltration.
  Oswestry Disability Index (ODI) will be calculated before and 1 month after procedure. This index (range 0 to 100) is used by clinicians and researchers to quantify disability for low back pain, with higher score indicating greater disability.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) score | 1 week
  Change in Oswestry Disability Index (ODI) score from baseline to 1 week after infiltration.
  Oswestry Disability Index (ODI) will be calculated before and 1 week after procedure. This index (range 0 to 100) is used by clinicians and researchers to quantify disability for low back pain, with higher score indicating greater disability.
Change in Visual Analog Scale (VAS) pain score from baseline to 1 week after infiltration | 1 week
  Pain will be evaluated by Visual Analog Scale (VAS) before and 1 week after infiltration. Visual Analog pain score (scale= 0 no pain; 10= worst pain imaginable)
Change in Visual Analog Scale (VAS) pain score from baseline to 1 month after infiltration | 1 month
  Pain will be evaluated by Visual Analog Scale (VAS) before and 1 month after infiltration.
  Visual Analog pain score (scale= 0 no pain; 10= worst pain imaginable)
Change in Duke Activity Status Index (DASI) from baseline to 1 week after infiltration | 1 week
  The Duke Activity Status Index (DASI) (range 0 to 58.2) will be calculated before and 1 week after procedure. This index is an assessment tool used to evaluate the possibility of carrying out daily activities, with higher scores indicating a higher functional capacity.
Change in Duke Activity Status Index (DASI) from baseline to 1 month after infiltration | 1 month
  The Duke Activity Status Index (DASI) (range 0 to 58.2) will be calculated before and 1 month after procedure. This index is an assessment tool used to evaluate the possibility of carrying out daily activities, with higher scores indicating a higher functional capacity.
Incidence of Adverse event (Hematoma, infection, intrathecal injection, spinal anesthesia) | 1 month
Hospital Anxiety and Depression Scale (HADS) | Before infiltration
  The Hospital Anxiety and Depression Scale (HADS) (range 0 to 21) will be calculated before procedure. (0-7 normal; 8-10 Borderline abnormal; 11-21 Abnormal)

CONTACTS AND LOCATIONS:
Overall Officials: Turgay Tuna, MD,PhD, Study Director — Erasme University Hospital; Marie-Laure Nisolle, MD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre; Panayota Kapessidou, MD,PhD, Study Chair — Centre Hospitalier Universitaire Saint Pierre
Locations (3):
- Belgium (3):
  - Hôpital de Braine l'Alleud Waterloo, Braine-l'Alleud
  - CHU Saint-Pierre, Brussels
  - Hôpital Erasme, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han SH, Park KD, Cho KR, Park Y. Ultrasound versus fluoroscopy-guided medial branch block for the treatment of lower lumbar facet joint pain: A retrospective comparative study. Medicine (Baltimore). 2017 Apr;96(16):e6655. doi: 10.1097/MD.0000000000006655. PMID 28422871
- [Background] Won HS, Yang M, Kim YD. Facet joint injections for management of low back pain: a clinically focused review. Anesth Pain Med (Seoul). 2020 Jan 31;15(1):8-18. doi: 10.17085/apm.2020.15.1.8. PMID 33329784
- [Background] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V. Lumbar facet joint nerve blocks in managing chronic facet joint pain: one-year follow-up of a randomized, double-blind controlled trial: Clinical Trial NCT00355914. Pain Physician. 2008 Mar-Apr;11(2):121-32. PMID 18354721
- [Background] Karkucak M, Batmaz I, Kerimoglu S, Ayar A. Comparison of clinical outcomes of ultrasonography-guided and blind local injections in facet syndrome: A 6-week randomized controlled trial. J Back Musculoskelet Rehabil. 2020;33(3):431-436. doi: 10.3233/BMR-181447. PMID 31524141
- [Background] Hurdle MF. Ultrasound-Guided Spinal Procedures for Pain: A Review. Phys Med Rehabil Clin N Am. 2016 Aug;27(3):673-86. doi: 10.1016/j.pmr.2016.04.011. PMID 27468672
- [Background] Ha DH, Shim DM, Kim TK, Kim YM, Choi SS. Comparison of ultrasonography- and fluoroscopy-guided facet joint block in the lumbar spine. Asian Spine J. 2010 Jun;4(1):15-22. doi: 10.4184/asj.2010.4.1.15. Epub 2010 Apr 26. PMID 20622950
- [Background] Kastler A, Kogl N, Gruber H, Skalla E, Loizides A. Lumbar medial branch cryoneurolysis under ultrasound guidance: initial report of five cases. Med Ultrason. 2020 Sep 5;22(3):293-298. doi: 10.11152/mu-2529. PMID 32898203
- [Background] Ye L, Wen C, Liu H. Ultrasound-guided versus low dose computed tomography scanning guidance for lumbar facet joint injections: same accuracy and efficiency. BMC Anesthesiol. 2018 Nov 7;18(1):160. doi: 10.1186/s12871-018-0620-7. PMID 30404599
- [Background] Kaye AD, Motejunas MW, Bonneval LA, Ehrhardt KP, Latimer DR, Trescot A, Wilson KE, Ibrahim IN, Cornett EM, Urman RD, Candido KD. Ultrasound practice for chronic pain procedures: A comprehensive review. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):465-486. doi: 10.1016/j.bpa.2019.07.001. Epub 2019 Jul 18. PMID 31791564
- [Background] Yun DH, Kim HS, Yoo SD, Kim DH, Chon JM, Choi SH, Hwang DG, Jung PK. Efficacy of ultrasonography-guided injections in patients with facet syndrome of the low lumbar spine. Ann Rehabil Med. 2012 Feb;36(1):66-71. doi: 10.5535/arm.2012.36.1.66. Epub 2012 Feb 29. PMID 22506237
- [Background] Boswell MV, Colson JD, Sehgal N, Dunbar EE, Epter R. A systematic review of therapeutic facet joint interventions in chronic spinal pain. Pain Physician. 2007 Jan;10(1):229-53. PMID 17256032
- [Background] Greher M, Kirchmair L, Enna B, Kovacs P, Gustorff B, Kapral S, Moriggl B. Ultrasound-guided lumbar facet nerve block: accuracy of a new technique confirmed by computed tomography. Anesthesiology. 2004 Nov;101(5):1195-200. doi: 10.1097/00000542-200411000-00020. PMID 15505456